CLINICAL TRIAL: NCT06521203
Title: Immediate Implant Placement in Sites With Chronic Periapical Lesions
Brief Title: Periapical Lesions and Immediate Implants
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Mehmet Ali Altay, Associate Professor, Akdeniz University
Other Study IDs: 20022019/188
Record Dates: First submitted 2024-07-17; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Dental Implant Failure Nos; Periapical Granuloma; Osseointegration Failure of Dental Implant
Keywords: Dental implant; Immediate dental implant; Osseointegrated implants; Osseointegration; Periapical granuloma; Tooth extraction
MeSH Terms: conditions — Periapical Granuloma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this case-control study is to evaluate the success and survival rates of dental implants immediately placed into extraction sites in the presence of periapical pathology.

The main questions it aims to answer are:

What were the survival and success rates of implants immediately placed into extraction sockets of teeth with chronic periodical lesions.

A retrospective analysis was performed based on the evaluation of certain clinical and radiographic parameters 12 months after prosthetic function of these implants.

DETAILED DESCRIPTION:
In 25 patients (13 men, 12 women), certain clinical and radiological parameters were retrospectively evaluated with particular interest in survival and success rates of the implants (total of 30 implants, 21 in the maxilla, 9 in the mandible) placed immediately to extraction sites of teeth with chronic periapical lesions. These parameters included mobility and the presence or absence of chronic pain, probing depth, gingival index, radiographic measurements of crestal bone loss on mesial and distal aspects of the implants.

ELIGIBILITY:
Inclusion Criteria:

* To have 1 or more teeth with a chronic periapical lesion that requiring extraction.
* The chronic periapical lesion should be determined as an asymptomatic periapical radiolucency with a diameter ranging between 4 and 8 mm.
* The patients undergoing tooth extraction must have been treated with an immediate implant placement procedure.
* At the time of extraction and implant placement, the neighboring teeth must have had healthy periodontal and periapical status.

Exclusion Criteria:

* Age younger than 18 years
* Any systemic disease or medication that might compromise osseointegration, bone or soft tissue healing
* Smoking
* Purulent exudate during the extraction
* Severe deficiency of soft and/or hard tissue in implant region
* Pregnancy
* Lactation
* History of chemotherapy or radiotherapy
* Severe parafunctional habits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The present study included patients, who underwent immediate implant placement following extraction of a tooth with periapical pathology.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Survival of the implants | Immediately after the implant placement and after 12 months of prosthesis function.
  Pain on palpation, percussion, or function (Yes/No) Implant mobility (Yes/No) Radiographic crestal bone loss (<4.0 mm) Absence of pain and mobility and crestal bone loss up to 4 mm were regarded as survive.
Success of the implants | Immediately after the implant placement and after 12 months of prosthesis function.
  Pain on palpation, percussion, or function (Yes/No) Implant mobility (Yes/No) Radiographic crestal bone loss (<2mm) Gingival index score (1-2-3) Probing depth (mm) Absence of pain and mobility, crestal bone loss <2mm, GI score less than 2, probing depth <5mm were regarded as success.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Adell R, Lekholm U, Rockler B, Branemark PI. A 15-year study of osseointegrated implants in the treatment of the edentulous jaw. Int J Oral Surg. 1981 Dec;10(6):387-416. doi: 10.1016/s0300-9785(81)80077-4. PMID 6809663
- [Background] Colak S, Demirsoy MS. Retrospective analysis of dental implants immediately placed in extraction sockets with periapical pathology: immediate implant placement in infected areas. BMC Oral Health. 2023 May 18;23(1):304. doi: 10.1186/s12903-023-02986-0. PMID 37208620
- [Background] Blanco J, Carral C, Argibay O, Linares A. Implant placement in fresh extraction sockets. Periodontol 2000. 2019 Feb;79(1):151-167. doi: 10.1111/prd.12253. PMID 30892772
- [Background] Koh RU, Rudek I, Wang HL. Immediate implant placement: positives and negatives. Implant Dent. 2010 Apr;19(2):98-108. doi: 10.1097/ID.0b013e3181d47eaf. PMID 20386212
- [Background] de Carvalho BC, de Carvalho EM, Consani RL. Flapless single-tooth immediate implant placement. Int J Oral Maxillofac Implants. 2013 May-Jun;28(3):783-9. doi: 10.11607/jomi.2140. PMID 23748309
- [Background] Gao Y, Luo D, Yuan M, Yang Y, Yang J. Immediate implant placement in single mandibular molar with chronic periapical periodontitis. J Stomatol Oral Maxillofac Surg. 2023 Dec;124(6S):101545. doi: 10.1016/j.jormas.2023.101545. Epub 2023 Jun 29. PMID 37390904
- [Background] Lang NP, Pun L, Lau KY, Li KY, Wong MC. A systematic review on survival and success rates of implants placed immediately into fresh extraction sockets after at least 1 year. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:39-66. doi: 10.1111/j.1600-0501.2011.02372.x. PMID 22211305
- [Background] Waasdorp JA, Evian CI, Mandracchia M. Immediate placement of implants into infected sites: a systematic review of the literature. J Periodontol. 2010 Jun;81(6):801-8. doi: 10.1902/jop.2010.090706. PMID 20192616
- [Background] Alsaadi G, Quirynen M, Komarek A, van Steenberghe D. Impact of local and systemic factors on the incidence of oral implant failures, up to abutment connection. J Clin Periodontol. 2007 Jul;34(7):610-7. doi: 10.1111/j.1600-051X.2007.01077.x. Epub 2007 Apr 13. PMID 17433044
- [Background] Truninger TC, Philipp AO, Siegenthaler DW, Roos M, Hammerle CH, Jung RE. A prospective, controlled clinical trial evaluating the clinical and radiological outcome after 3 years of immediately placed implants in sockets exhibiting periapical pathology. Clin Oral Implants Res. 2011 Jan;22(1):20-7. doi: 10.1111/j.1600-0501.2010.01973.x. PMID 20678132
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. BMJ. 2007 Oct 20;335(7624):806-8. doi: 10.1136/bmj.39335.541782.AD. PMID 17947786
- [Background] Misch CE, Perel ML, Wang HL, Sammartino G, Galindo-Moreno P, Trisi P, Steigmann M, Rebaudi A, Palti A, Pikos MA, Schwartz-Arad D, Choukroun J, Gutierrez-Perez JL, Marenzi G, Valavanis DK. Implant success, survival, and failure: the International Congress of Oral Implantologists (ICOI) Pisa Consensus Conference. Implant Dent. 2008 Mar;17(1):5-15. doi: 10.1097/ID.0b013e3181676059. PMID 18332753
- [Background] Ainamo J, Bay I. Problems and proposals for recording gingivitis and plaque. Int Dent J. 1975 Dec;25(4):229-35. PMID 1058834
- [Background] Suzuki JB, Misch CE. Periodontal and maintenance complications. In: Resnik RR, Misch CE, eds. Misch's Avoiding Complications in Oral Implantology. Elsevier; 2017:771-826.
- [Background] Maheshwari R, Punia V, Khandelwal M, Sharma V, Malot S, Porwal A. Implant failure and management: A review. IJADS. 2018;4:293-8.
- [Background] Koo TK, Li MY. A Guideline of Selecting and Reporting Intraclass Correlation Coefficients for Reliability Research. J Chiropr Med. 2016 Jun;15(2):155-63. doi: 10.1016/j.jcm.2016.02.012. Epub 2016 Mar 31. PMID 27330520
- [Background] Alvarez-Camino JC, Valmaseda-Castellon E, Gay-Escoda C. Immediate implants placed in fresh sockets associated to periapical infectious processes. A systematic review. Med Oral Patol Oral Cir Bucal. 2013 Sep 1;18(5):e780-5. doi: 10.4317/medoral.18942. PMID 23722139
- [Background] Lindeboom JA, Tjiook Y, Kroon FH. Immediate placement of implants in periapical infected sites: a prospective randomized study in 50 patients. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Jun;101(6):705-10. doi: 10.1016/j.tripleo.2005.08.022. Epub 2006 Mar 22. PMID 16731387
- [Background] Lazzara RJ. Immediate implant placement into extraction sites: surgical and restorative advantages. Int J Periodontics Restorative Dent. 1989;9(5):332-43. No abstract available. PMID 2640210
- [Background] Novaes AB Jr, Vidigal Junior GM, Novaes AB, Grisi MF, Polloni S, Rosa A. Immediate implants placed into infected sites: a histomorphometric study in dogs. Int J Oral Maxillofac Implants. 1998 May-Jun;13(3):422-7. PMID 9638015
- [Background] Chang SW, Shin SY, Hong JR, Yang SM, Yoo HM, Park DS, Oh TS, Kye SB. Immediate implant placement into infected and noninfected extraction sockets: a pilot study. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2009 Feb;107(2):197-203. doi: 10.1016/j.tripleo.2008.06.003. Epub 2008 Aug 28. PMID 18755614
- [Background] Khademi A, Shadmehr E, Ajami M, Rismanchian M, Razavi SM. Histologic and histomorphometric assessment of implants and periapical tissues when placed in the sockets of extracted teeth, teeth with periapical lesions, and healed lesions: a canine study. J Oral Implantol. 2013 Dec;39(6):709-13. doi: 10.1563/AAID-JOI-D-11-00137. Epub 2011 Nov 21. PMID 22103780
- [Background] Casap N, Zeltser C, Wexler A, Tarazi E, Zeltser R. Immediate placement of dental implants into debrided infected dentoalveolar sockets. J Oral Maxillofac Surg. 2007 Mar;65(3):384-92. doi: 10.1016/j.joms.2006.02.031. PMID 17307582
- [Background] Karoussis IK, Salvi GE, Heitz-Mayfield LJ, Bragger U, Hammerle CH, Lang NP. Long-term implant prognosis in patients with and without a history of chronic periodontitis: a 10-year prospective cohort study of the ITI Dental Implant System. Clin Oral Implants Res. 2003 Jun;14(3):329-39. doi: 10.1034/j.1600-0501.000.00934.x. PMID 12755783
- [Background] Esposito M, Grusovin MG, Polyzos IP, Felice P, Worthington HV. Timing of implant placement after tooth extraction: immediate, immediate-delayed or delayed implants? A Cochrane systematic review. Eur J Oral Implantol. 2010 Autumn;3(3):189-205. PMID 20847990
- [Background] Lee CT, Chuang SK, Stoupel J. Survival analysis and other clinical outcomes of immediate implant placement in sites with periapical lesions: systematic review. Int J Oral Maxillofac Implants. 2015 Mar-Apr;30(2):268-78. doi: 10.11607/jomi.3619. PMID 25830386
- [Background] Fugazzotto PA. A retrospective analysis of implants immediately placed in sites with and without periapical pathology in sixty-four patients. J Periodontol. 2012 Feb;83(2):182-6. doi: 10.1902/jop.2011.110016. Epub 2011 May 31. PMID 21627462
- [Background] Fugazzotto P. A retrospective analysis of immediately placed implants in 418 sites exhibiting periapical pathology: results and clinical considerations. Int J Oral Maxillofac Implants. 2012 Jan-Feb;27(1):194-202. PMID 22299097
- [Background] Montoya-Salazar V, Castillo-Oyague R, Torres-Sanchez C, Lynch CD, Gutierrez-Perez JL, Torres-Lagares D. Outcome of single immediate implants placed in post-extraction infected and non-infected sites, restored with cemented crowns: a 3-year prospective study. J Dent. 2014 Jun;42(6):645-52. doi: 10.1016/j.jdent.2014.03.008. Epub 2014 Mar 24. PMID 24675527
- [Background] Novaes AB Jr, Novaes AB. Immediate implants placed into infected sites: a clinical report. Int J Oral Maxillofac Implants. 1995 Sep-Oct;10(5):609-13. PMID 7591007
- [Background] Siegenthaler DW, Jung RE, Holderegger C, Roos M, Hammerle CH. Replacement of teeth exhibiting periapical pathology by immediate implants: a prospective, controlled clinical trial. Clin Oral Implants Res. 2007 Dec;18(6):727-37. doi: 10.1111/j.1600-0501.2007.01411.x. Epub 2007 Sep 20. PMID 17888019
- [Background] Villa R, Rangert B. Early loading of interforaminal implants immediately installed after extraction of teeth presenting endodontic and periodontal lesions. Clin Implant Dent Relat Res. 2005;7 Suppl 1:S28-35. doi: 10.1111/j.1708-8208.2005.tb00072.x. PMID 16137085
- [Background] Del Fabbro M, Boggian C, Taschieri S. Immediate implant placement into fresh extraction sites with chronic periapical pathologic features combined with plasma rich in growth factors: preliminary results of single-cohort study. J Oral Maxillofac Surg. 2009 Nov;67(11):2476-84. doi: 10.1016/j.joms.2009.04.063. PMID 19837321